CLINICAL TRIAL: NCT03155854
Title: The Effects of Prophylactic Limited Palmar Fasciectomy on Surgical Outcomes and Scarring for Dupuytren's Contracture Patients With Pretendinous Cord - Prospective Randomized Clinical Study (Pilot)
Brief Title: The Effects of Prophylactic Limited Palmar Fasciectomy on Surgical Outcomes and Scarring
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Sanjeev (Sanj) Kakar, M.D., M.B.A., Professor of Orthopedics,, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-008280
Record Dates: First submitted 2016-10-07; First posted 2017-05-16 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Dupuytren Contracture
MeSH Terms: conditions — Dupuytren Contracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pretendinous cord excision (Active Comparator): Patients will undergo either a targeted palmar fasciectomy procedure in which the involved Dupuytren's fascia will be excised
  Interventions: Procedure: Pretendinous cord excision
- Division/manipulation of the cord (Active Comparator): patients will undergo either a targeted palmar fasciectomy procedure in which the involved Dupuytren's fascia will be incised.
  Interventions: Procedure: Division/manipulation of the cord

INTERVENTIONS:
Procedure: Pretendinous cord excision — The cord/palmar fascia will be excised during surgery.
  Arms: Pretendinous cord excision
Procedure: Division/manipulation of the cord — The pretendinous cord will be divided and incised during surgery.
  Arms: Division/manipulation of the cord

SUMMARY:
Research is instrumental for improving medical care and the patient experience. Finding new surgical techniques can create better outcomes and minimize recovery time and complications for patients. Some patients undergoing trigger finger surgery with a pre-existing Dupuytren's cord may develop a thickened surgical scar after surgery, which can cause discomfort, difficulty with moving or using, and other complications in the affected finger(s) or hand. The investigator is investigating a surgical technique to minimize these potential complications and scarring after surgery.

Subjects are being asked to take part in this research study because they have been diagnosed with trigger finger and pretendinous Dupuytren's cord and have decided to undergo surgery rather than try medical treatment.

DETAILED DESCRIPTION:
Patients who have surgery for trigger finger with a thickened overlying Dupuytren's cord are at risk for complications including but not limited to scarring, adhesions, stiffness, injury to underlying structures such as blood vessels, tendons and nerves, loss of motion, pain, bowstringing, and recurrent triggering or contracture. They have been shown to have higher risk for these complications including a thickened scar response. The cause for this is not fully understood, but it could be because the pretendinous cord was cut and not removed. By cutting and not removing this pretendinous cord, this may cause extra scarring that may lead to a thicker palmar scar that may become symptomatic. This study will investigate a different surgical method for relieving the tension caused by a pretendinous cord and whether it reduces complications and scarring.

ELIGIBILITY:
Inclusion Criteria:

* Potential candidates for the study will be selected based upon clinical diagnosis of trigger finger with co-existing pretendinous cord. All potential subjects will have either failed non operative treatment or elected surgical treatment.

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Scar Progression as measured by the Vancouver Scar Scale | baseline, up to 1 year
  The Vancouver Scar Scale assesses 4 variables: vascularity, height/thickness, pliability, and pigmentation. Patient perception of his or her respective scars is not factored in to the overall score. The scores can range from 0 (normal) to 13 (severe scarring).
Change in Scar Progression as measured by the Patient and Observer Scar Assessment Scale | baseline, up to 1 year
  The Patient and Observer Scar Assessment Scale consists of two parts: a Patient Scale and an Observer Scale. Both scales contain seven items that are scored numerically on a 10-step scale. Together they make up the 'Total Score' of the Patient and Observer Scale. The total score can range from 14 (normal) to 140 (worst scar imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Sanjeev Kakar, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials